CLINICAL TRIAL: NCT05604066
Title: Magnetic Resonance Elastography of Myofascial Pain Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Ziying Yin, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-007647; R61AT012185 (NIH)
Record Dates: First submitted 2022-10-24; First posted 2022-11-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Myofascial Pain
Keywords: Magnetic Resonance Imaging (MRI); Magnetic Resonance Elastography (MRE)
MeSH Terms: interventions — Magnetic Resonance Imaging; Elasticity Imaging Techniques

STUDY DESIGN:
Intervention Model Description: This is a two-phase NIH-awarded study. The first R61 phase (currently awarded) is an observational study with one control group and one patient group. The second R33 phase is a pilot clinical trial, which will be awarded by the end of the R61 phase. The study design provided here is for R61 only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with myofascial-related pain diseases (Experimental): Subjects diagnosed with myofascial-related pain disease will receive the research MRI imaging including MR elastography and MRI structural imaging.
  Interventions: Diagnostic Test: Magnetic Resonance (MR) Elastography; Diagnostic Test: MRI structural imaging
- Healthy controls without myofascial-related pain diseases (Experimental): Subjects without myofascial-related pain disease will receive the research MRI imaging including MR elastography and MRI structural imaging.
  Interventions: Diagnostic Test: Magnetic Resonance (MR) Elastography; Diagnostic Test: MRI structural imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance (MR) Elastography — Magnetic resonance imaging (MRI) imaging technique that creates a visual map (Elastogram) to show the stiffness of body tissues
  Other Names: MRE
Diagnostic Test: MRI structural imaging — MRI structural imaging will be done at the same time as MR elastography.
  Other Names: MRI

SUMMARY:
The purpose of this research study is to use a new imaging technique called Magnetic Resonance (MR) Elastography to create new imaging parameters to measure the mechanical properties of myofascial tissues that can be used to assess the impaired myofascial interface in myofascial pain syndrome (MPS).

DETAILED DESCRIPTION:
This is observational research that aims to develop an MRI-based imaging technique (MRE) to quantitatively assess the myofascial tissue properties in healthy subjects and patients with relevant pain conditions. Healthy volunteers and patients with MPS will be recruited to undergo MRI along with MR elastography.

ELIGIBILITY:
Healthy Volunteer Inclusion Criteria:

* Absence of a history of chronic pain in the targeted anatomical location (i.e., lower back and low extremities) that had limited activities of daily living or work
* A numerical current pain index of less than 0.5 (on a 10-point Visual Analog Scale)
* Able to understand the goal of the project and give informed consent.

Healthy Volunteer Exclusion Criteria:

* Pregnancy or breastfeeding
* Any contraindication to an MRI exam
* Previous severe/acute back or low extremity injury (including fracture)
* Previous back or low extremity surgery
* Back and lower limb deformities
* Inability to provide consent.

Myofascial-Related Pain Patient Inclusion Criteria:

* A history of chronic low back or leg pain (the targeted location will be determined based on the findings in Aim 1) for at least 3 months. (Measured by patient history and physical exam)
* A palpable taut band or nodule within the skeletal muscle
* Hypersensitive tender spot within the taut band
* Recognition of current pain complaint by pressure on the tender nodule/taut band
* Painful limit to the full stretch range of motion

Myofascial-Related Pain Patient Exclusion Criteria:

* Pregnancy or breastfeeding
* Any contraindication to an MRI exam
* Previous therapy in the area to be treated within 6 months
* Previous severe back or low extremity injury (including fracture) or surgery
* Any neurological conditions or active systemic disease (e.g. diabetes, peripheral vascular disease, cancer, rheumatoid arthritis) that impaired sensation/pain perception
* Severe osteoarthritis
* Skin injuries in the area to be treated
* Inability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The fascia plane mobility assessed by MR Elastography-based normalized octahedral shear strain (NOSS) measurements | baseline measures through the study completion (3 years)
  In response to an external shear force, the fascial layers that surround and separate muscles can deform or slide relative to each other, depending on the fascial plane's mobility. An adhesive interface that experiences a shear force will exhibit shear displacement continuity (i.e., small shear strain) across the interface, while a nonadhesive interface may slip rather than deform, which causes a discontinuity in displacement (i.e., large shear strain). For the targeted fascia plane in low back and legs, the normalized octahedral shear strain (NOSS) will be computed from the shear displacement data measured from MRE to assess the fascia plane mobility. The primary outcome measure is the difference in the fascia plane mobility on MR elastography between patients with myofascial-related pain diseases and healthy controls without myofascial-related pain diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Ziying Yin, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials